CLINICAL TRIAL: NCT07358078
Title: DemonsTTRate: A Global, Observational, Multicenter, Long-term Study of Patients With Transthyretin-Mediated Amyloidosis With Cardiomyopathy in a Real-World Setting
Brief Title: DemonsTTRate: A Global, Observational, Multicenter, Long-term Study of Patients With ATTR-CM in a Real-World Setting
Acronym: DemonsTTRate
Status: Recruiting | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTRSC02-008
Record Dates: First submitted 2025-11-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Amyloidosis With Cardiomyopathy
Keywords: ATTR-CM; Transthyretin; Amyloidosis; ATTR; Cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with ATTR-CM: Patients with ATTR-CM.

SUMMARY:
The purpose of this study is to:

* Describe the clinical characteristics of adult patients with transthyretin-mediated amyloidosis with cardiomyopathy (ATTR-CM) treated with vutrisiran in routine clinical care
* Describe treatment patterns of adult patients with ATTR-CM treated with vutrisiran in routine clinical care
* Assess health-related quality of life (HRQOL) in adult patients with ATTR-CM treated with vutrisiran in routine clinical care
* Assess healthcare resource use (HCRU) in adult patients with ATTR-CM treated with vutrisiran in routine clinical care Compare the long-term effectiveness of vutrisiran versus other approved ATTR-CM treatments in routine clinical care

DETAILED DESCRIPTION:
Each site will invite all eligible patients to participate. Patients will be followed for up to 5 years or until patient withdrawal of consent, loss to follow-up, death, or the end of the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of ATTR-CM
* Is initiating treatment with vutrisiran or another approved ATTR-CM therapy

Exclusion Criteria:

* Is enrolled in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients with ATTR-CM who, at enrollment, are either initiating treatment with vutrisiran or are initiating treatment with another approved ATTR-CM therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2030-10-23 (Estimated); Study Completion 2030-10-23 (Estimated)

PRIMARY OUTCOMES:
New York Heart Association (NYHA) Class | From time of ATTR-CM diagnosis up to 5 years
  The NYHA functional classification categorizes the severity of heart failure. Patients are classified in 1 of 4 categories based on their physical limitations, as follows:
  * Class I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or shortness of breath.
  * Class II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  * Class III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  * Class IV Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Outpatient Diuretic Intensification | From time of enrollment for up to 5 years
  The clinician-reported outcome of ODI, which measures any post-diagnosis initiation or increase in the dose of loop diuretics, may help identify patients with ATTR-CM who are at an increased risk for adverse outcomes. ODI, a marker to monitor disease progression and/or worsening heart failure, is associated with a higher risk of all-cause mortality, cardiovascular hospitalizations, and urgent heart failure visits. Clinicians monitor ODI to help manage patients with ATTR-CM.
Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) Total Score | From time of enrollment (if available) or ATTR-CM diagnosis up to 5 years
  Norfolk-QoL-DN: The Norfolk QOL-DN questionnaire is a standardized 35-item patient-reported outcomes measure that assesses 6 domains: physical function, large-fiber neuropathy, activities of daily living, symptoms, small-fiber neuropathy, and autonomic neuropathy. The total score ranges from -4 points (best possible quality of life) to 136 points (worst possible quality of life).
Kansas City Cardiomyopathy Questionnaire (KCCQ) | From time of enrollment (if available) or ATTR-CM diagnosis up to 5 years
  The KCCQ is a 23-item self-administered questionnaire developed to independently measure the patient's perception of health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life within a 2-week recall period. The KCCQ quantifies 6 domains (symptoms, physical function, quality of life, social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and overall summary [OS] scores).
Patient Global Impressions - Change (PGI-C) | From time of enrollment (if available) or ATTR-CM diagnosis up to 5 years
  The PGI-C is a 7-point numerical rating scale where 1 indicates "very much improved" and 7 indicates "very much worse."
Patient Global Impressions - Severity (PGI-S); | From time of enrollment (if available) or ATTR-CM diagnosis up to 5 years
  The PGI-S is a 7-point numerical rating scale where 1 indicates "very much improved" and 7 indicates "very much worse."
Treatment Satisfaction Questionnaire for Medication version 9 (TSQM-9) | From time of enrollment (if available) or ATTR-CM diagnosis up to 5 years
  TSQM-9 is a 9-item general instrument that measures the major dimensions of satisfaction with a medication. The questionnaire consists of 3 domains: effectiveness, convenience and side effects. The scores of each domain range from 0 to 100 with higher scores representing higher satisfaction on that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals Inc
Locations (1):
- Clinical Trial Site, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No